CLINICAL TRIAL: NCT03745872
Title: SunSmart Intervention in Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-0667.cc
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Melanoma
Keywords: Sunscreen; Sun Exposure; Behaviors; Baseline Assessments; Follow-up Assessments; Knowledge
MeSH Terms: conditions — Melanoma; Behavior

STUDY DESIGN:
Intervention Model Description: All students who participate in this study will be given a pre test, instruction regarding sun exposure and a post test to determine their sun exposure behaviors and knowledge of sun exposure risks.
Masking Description: Participant names will be written on pre and post test to enable matching purposes, but once this has been completed, only the study ID will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testing (Experimental): This is a preventative study model. All students who choose to participate will receive a pre and post test regarding their sun exposure behaviors and knowledge on sun exposure risk.
  Interventions: Behavioral: Knowledge Assessment

INTERVENTIONS:
Behavioral: Knowledge Assessment — Students participating in this study will receive a pre test, instruction regarding sun safety, and a post test.

SUMMARY:
A prevention study to improve sun exposure behaviors in children after an educational classroom-based intervention.

DETAILED DESCRIPTION:
This study aims to demonstrate that learning about sun exposure using a more classroom-based intervention will motivate classroom students to reduce exposure at a critical life period and will create lifetime learned sun exposure behaviors. Students' sun exposure behaviors will be assessed prior to the educational intervention. The educational intervention consists of three educational sessions and one lab lesson. At the conclusion of the intervention, students' sun exposure behaviors will be assessed again via a post-intervention questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Any children between grades 4 and 8 enrolled in one of the participating schools.

Exclusion Criteria:

* No exclusions, but children or their parents may opt out of participating.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Sun Exposure Knowledge | From the administration of the questionnaire to the end of the followup questionnaire, up to 3 years
  Determining children's knowledge of sun exposure risk through a self-completed questionnaire
Sun Exposure Attitudes | From the administration of the questionnaire to the end of the followup questionnaire, up to 3 years
  Determining children's attitude toward sun exposure through a self-completed questionnaire
Sun Exposure Behavior | From the administration of the questionnaire to the end of the followup questionnaire, up to 3 years
  Determining children's behavior toward sun exposure through a self-completed questionnaire

SECONDARY OUTCOMES:
Mediators of Program Effects: Attitudes | During the followup questionnaire, which is given 3 to 4 weeks post intervention, up to three years
  Assessing children's attitude toward sun exposure through a self-completed questionnaire
Mediators of Program Effects: Norms | During the followup questionnaire, which is given 3 to 4 weeks post intervention, up to three years
  Determining children's understanding of social norms regarding tanning and sun protection through a self-completed questionnaire
Mediators of Program Effects: Personal Agency | During the followup questionnaire, which is given 3 to 4 weeks post intervention, up to three years
  Determining children's understanding of behavioral control regarding sun protection through a self-completed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Evelinn Borrayo, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States